CLINICAL TRIAL: NCT02126839
Title: A Three-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Chronic-Dose Safety and Efficacy Study of Albuterol Multi-Dose Dry Powder Inhaler (MDPI) Relative to Placebo in Pediatric Asthmatics
Brief Title: A Chronic-Dose Safety and Efficacy Study of Albuterol Multi-Dose Dry Powder Inhaler in Pediatric Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABS-AS-303
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo MDPI QID (Placebo Comparator): Placebo multidose dry powder inhaler (MDPI) administered as 2 inhalations QID (at approximately 7:00 AM, 12 noon, 5:00 PM, and bedtime) for 3 weeks.
  Interventions: Drug: Placebo; Drug: ProAir HFA inhaler
- Albuterol MDPI 180 mcg QID (Experimental): Albuterol multidose dry powder inhaler (MDPI) 90 mcg/inhalation administered as 2 inhalations QID (at approximately 7:00 AM, 12 noon, 5:00 PM, and bedtime) for a total daily dose of 720 mcgs for 3 weeks.
  Interventions: Drug: Albuterol MDPI; Drug: ProAir HFA inhaler

INTERVENTIONS:
Drug: Albuterol MDPI — 90 mcg/actuation of the multidose dry powder inhaler (MDPI).
  Other Names: Spiromax®
  Arms: Albuterol MDPI 180 mcg QID
Drug: Placebo — Matching Placebo delivered via a multidose dry powder inhaler (MDPI).
  Arms: Placebo MDPI QID
Drug: ProAir HFA inhaler — Rescue medication, ProAir hydrofluoroalkane (HFA) inhaler, was dispensed at the run-in visit for the relief of asthma symptoms to be administered as needed.
  Other Names: albuterol

SUMMARY:
The study is to evaluate the chronic-dose efficacy and the safety of Albuterol MDPI compared to placebo in pediatric participants with asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent signed and dated by the patient and/or parent/caregiver/legal guardian (as appropriate) before conducting any study related procedure
2. Male or premenarchal female 4-11 years of age, inclusive, as of the screening visit (SV)
3. Has a documented physician diagnosis of asthma per the EPR-3 Guidelines of a minimum of 6 months duration that has been stable for at least 4 weeks prior to the SV
4. Has the ability to perform spirometry reproducibly consistent with ATS guidelines and protocol-specific guidelines
5. Has FEV1 50-95% predicted for age, height and gender at the SV following a minimum 6-hour period without β2-agonist use. (Note: Predicted values of 49.50-49.99% may be rounded up to 50% and values of 95.01-95.49% may be rounded down to 95%.)
6. Demonstrated reversible bronchoconstriction as verified by a 15% or greater increase in baseline FEV1 within 30 minutes following inhalation of 180 mcg of albuterol. (Note: Reversibility values of 14.50-14.99% may be rounded up to 15%.)
7. Is maintained on low-dose inhaled corticosteroids (ICS, less than or equal to 200 mcg of fluticasone propionate per day or equivalent), leukotriene modifiers (LTM), or inhaled cromones, and/or on short-acting β2-agonists (SABA); as needed SABA alone is acceptable. The ICS, LTM, and cromone doses must have been stable for at least 4 weeks prior to the SV and should be maintained for the duration of the study
8. Can self-perform peak expiratory flow rate (PEF) measurements with a handheld peak flow meter
9. Can tolerate the withdrawal of applicable medications for qualification at screening
10. Otherwise in general good health, defined as free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the trial, and with a clinically acceptable 6-month medical history, physical examination, 12-lead electrocardiogram (ECG), and vital signs
11. Parents consenting are capable of understanding the requirements, risks and benefits of study participation, and, as judged by the investigator, capable of giving informed consent and being compliant with all study requirements (eg, visits, record-keeping)
12. The patient is able to correctly use the MDPI device, either alone or with assistance by a parent/guardian.

Exclusion Criteria

1. Known hypersensitivity to albuterol or any of the excipients in the inhaler formulations (eg, lactose, ethanol)
2. Participation (receiving study medication) in any investigational drug trial within the 30 days preceding the SV or planned participation in another investigational drug trial at any time during this trial
3. History of severe milk protein allergy
4. History of a respiratory infection or disorder (including, but not limited to bronchitis, pneumonia, acute or chronic sinusitis, otitis media, influenza) that has not resolved within 4 weeks preceding the SV
5. Any asthma exacerbation requiring oral corticosteroids within 3 months of the SV. A patient must not have had any hospitalization for asthma within 6 months prior to the SV.
6. Initiation of immunotherapy during the study period or dose escalation during the study period. Patients being treated with immunotherapy prior to the SV must be using a stable (maintenance) dose (90 days or more) to be considered for inclusion.
7. History of life-threatening asthma that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest, or hypoxic seizures
8. Use of any prohibited concomitant medications within the washout prescribed per protocol prior to study visits
9. Use of any medication for asthma or allergic rhinitis that is prohibited per the protocol as described in the protocol
10. The dosage of any required LTM, ICS, or inhaled cromones, has not been stable for at least 4 weeks. Intranasal corticosteroid and/or cromones have not been stable for at least two weeks prior to the SV. Allowed corticosteroid, LTM, and cromone asthma and allergy medications should be continued at the same doses during the conduct of the study.
11. Presence of any non-asthmatic acute or chronic condition, including but not limited to bronchitis, emphysema, active tuberculosis, bronchiectasis, cystic fibrosis, clinically significant cardiovascular disease (including but not limited to cardiac arrhythmias and uncontrolled hypertension), clinically significant hepatic, renal, or endocrine dysfunction, stroke, uncontrolled diabetes mellitus, hyperthyroidism, convulsive disorder, and malignancy other than basal cell carcinoma. Significant is defined as any condition that, in the opinion of the investigator, would put the safety of the patient at risk through participation, or which could affect the safety or efficacy analyses
12. Any other medical or psychological condition that in the investigator's opinion should preclude study enrollment
13. Previous participation (received MDPI study medication) in an Albuterol MDPI study
14. Study participation by clinical investigator site employees and/or their immediate relatives
15. Study participation by related or non-related individuals living in the same household, ie, only one subject per household may participate in the study at the same time.
16. Require continuous treatment with β-blockers, MAO inhibitors, tricyclic antidepressants, anticholinergics, and/or systemic corticosteroids
17. Treated with oral or injectable corticosteroids within the 6 weeks prior to SV
18. Hospitalization for acute asthma exacerbation >2 times in 12 months prior to screening and/or received emergency room treatment other than nebulized albuterol or been hospitalized for asthma exacerbations within 6 months prior to SV

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (52):
- United States (51):
  - Teva Investigational Site 12496, Birmingham, Alabama
  - Teva Investigational Site 12500, Mobile, Alabama
  - Teva Investigational Site 12481, Little Rock, Alaska
  - Teva Investigational Site 12515, Anaheim, California
  - Teva Investigational Site 12505, Costa Mesa, California
  - Teva Investigational Site 12476, Huntington Beach, California
  - Teva Investigational Site 12519, Los Angeles, California
  - Teva Investigational Site 12484, Mission Viejo, California
  - Teva Investigational Site 12510, Riverside, California
  - Teva Investigational Site 12483, Rolling Hills Estates, California
  - Teva Investigational Site 12511, Sacramento, California
  - Teva Investigational Site 12485, Stockton, California
  - Teva Investigational Site 12512, Centennial, Colorado
  - Teva Investigational Site 12522, Gainesville, Florida
  - Teva Investigational Site 12535, Hollywood, Florida
  - Teva Investigational Site 12526, Miami, Florida
  - Teva Investigational Site 12516, Orlando, Florida
  - Teva Investigational Site 12517, Tamarac, Florida
  - Teva Investigational Site 12527, Vero Beach, Florida
  - Teva Investigational Site 12513, Winter Park, Florida
  - Teva Investigational Site 12486, Gainesville, Georgia
  - Teva Investigational Site 12497, Lawrenceville, Georgia
  - Teva Investigational Site 12480, Savannah, Georgia
  - Teva Investigational Site 12508, Shiloh, Illinois
  - Teva Investigational Site 12518, Iowa City, Iowa
  - Teva Investigational Site 12523, Covington, Louisiana
  - Teva Investigational Site 12495, Warrensburg, Missouri
  - Teva Investigational Site 12509, Northfield, New Jersey
  - Teva Investigational Site 12524, Brooklyn, New York
  - Teva Investigational Site 12473, Raleigh, North Carolina
  - Teva Investigational Site 12477, Cincinnati, Ohio
  - Teva Investigational Site 12525, Cleveland, Ohio
  - Teva Investigational Site 12502, Middleburg Heights, Ohio
  - Teva Investigational Site 12478, Oklahoma City, Oklahoma
  - Teva Investigational Site 12487, Oklahoma City, Oklahoma
  - Teva Investigational Site 12506, Oklahoma City, Oklahoma
  - Teva Investigational Site 12492, Tulsa, Oklahoma
  - Teva Investigational Site 12507, Gresham, Oregon
  - Teva Investigational Site 12501, Normal Square, Pennsylvania
  - Teva Investigational Site 12493, Pittsburgh, Pennsylvania
  - Teva Investigational Site 12488, Upland, Pennsylvania
  - Teva Investigational Site 12514, Greenville, South Carolina
  - Teva Investigational Site 12474, Orangeburg, South Carolina
  - Teva Investigational Site 12479, Spartanburg, South Carolina
  - Teva Investigational Site 12489, Boerne, Texas
  - Teva Investigational Site 12475, Waco, Texas
  - Teva Investigational Site 12491, Burke, Virginia
  - Teva Investigational Site 12504, Charlottesville, Virginia
  - Teva Investigational Site 12482, Richmond, Virginia
  - Teva Investigational Site 12498, Richmond, Virginia
  - Teva Investigational Site 12490, Spokane, Washington
- Teva Investigational Site 12533, Papillion, NE, Thailand

REFERENCES:
- [Derived] Ratnayake A, Taveras H, Iverson H, Shore P. Pharmacokinetics and pharmacodynamics of albuterol multidose dry powder inhaler and albuterol hydrofluoroalkane in children with asthma. Allergy Asthma Proc. 2016 Sep;37(5):370-5. doi: 10.2500/aap.2016.37.3985. Epub 2016 Aug 12. PMID 27523719

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The run-in period (days -14 to Day -1) was conducted in a single blind manner with respect to the Placebo MDPI treatment (2 inhalations QID at approximately 7:00 AM, 12:00 PM, 5:00 PM, and bedtime), so that the patient did not know which treatment was administered.
Period: Overall Study
Arm/Group | Placebo MDPI QID | Albuterol MDPI 180 mcg QID
Started | 92 | 94
Safety Population | 92 | 93
Full Analysis Set | 92 | 92
Completed | 82 | 80
Not Completed | 10 | 14
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal by parent/guardian | 1 | 0
Not completed — Protocol Violation | 2 | 3
Not completed — Sponsor request | 0 | 1
Not completed — Lost to Follow-up | 1 | 4
Not completed — Other | 5 | 5

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo MDPI QID | Albuterol MDPI 180 mcg QID | Total
Number analyzed (Participants) | 92 | 94 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (1.83) | 8.3 (1.69) | 8.4 (1.76)
Age, Customized [Number; unit: participants]
  4-7 years | 23 | 30 | 53
  8-11 years | 69 | 64 | 133
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 42 | 79
  Male | 55 | 52 | 107
Race/Ethnicity, Customized [Number; unit: participants]
  White | 41 | 40 | 81
  Black | 48 | 52 | 100
  American Indian or Alaskan Native | 0 | 1 | 1
  Pacific Islander | 0 | 1 | 1
  Other | 3 | 0 | 3
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 11 | 14 | 25
  Not Hispanic or Latino | 81 | 80 | 161
Weight [Mean (Standard Deviation); unit: kg] | 37.2 (13.42) | 36.1 (13.46) | 36.7 (13.42)
Height [Mean (Standard Deviation); unit: cm] | 136.9 (12.67) | 135.2 (11.59) | 136.0 (12.13)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 19.5 (4.96) | 19.4 (5.34) | 19.4 (5.14)
Screening FEV1 [Mean (Standard Deviation); unit: liters] — FEV1 = forced expiratory volume in 1 second
  liters | 1.69 (0.44) | 1.64 (0.35) | 1.66 (0.39)
Screening PPFEV1 [Mean (Standard Deviation); unit: percent of predicted FEV1] — PPFEV1 = percent-predicted forced expiratory volume in 1 second
  percent of predicted FEV1 | 87.5 (11.46) | 89.0 (12.35) | 88.3 (11.91)
Qualifying Airway Reversibility [Mean (Standard Deviation); unit: percentage increase from baseline FEV1] — For a patient to be eligible for study enrollment, a minimum of 15% increase from the baseline FEV1 must be demonstrated after receiving 180 mcg of albuterol, administered as 2 actuations 1 minute apart.
  percentage increase from baseline FEV1 | 22.0 (8.14) | 22.9 (8.19) | 22.4 (8.16)

OUTCOME MEASURES:

1. Primary Outcome: Baseline Adjusted Percent Predicted Forced Expiratory Volume In 1 Second (FEV1) Area Under The Concentration Time Curve Up From Time Zero up to 6 Hours (AUC0-6) Over 3 Weeks
Description: Following measurement of the baseline FEV1 and dose administration on Days 1 and 22, FEV1 values (highest of 3 acceptable maneuvers) will be obtained at 5 (±2), 15 (±5), 30 (±5), 45 (±5), 60 (±10), 120 (±10), 240 (±10), and 360 (±10) minutes after the completion of dosing. Predicted FEV1 values were computed and adjusted for age, height, and gender according to Eigen et al (Eigen et al 2001) for participants 4 to 5 years of age and to Quanjer et al (Quanjer et al 1995) for participants aged 6 to 11 years using ATS criteria (American Thoracic Society/European Respiratory Society Statement 2007).
Time Frame: 30 ±5 and 5 ±2 minutes prior to dosing, and at 5 ±2, 15 ±5, 30 ±5, 45 ±5, 60 ±10, 120 ±10, 240 ±10, and 360 ±10 minutes after completion of dosing on Days 1 and 22
Population: The full analysis set (FAS) includes all participants in the ITT population who receive at least 1 dose of study medication and have at least 1 postbaseline assessment of the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: % predicted FEV1/hour
Arm/Group | Placebo MDPI QID | Albuterol MDPI 180 mcg QID
Number analyzed (Participants) | 92 | 92
% predicted FEV1/hour | 18.71 (3.190) | 43.73 (3.200)
Statistical Analysis 1: Comparison: Placebo MDPI QID vs Albuterol MDPI 180 mcg QID; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures analysis; Fixed effects of treatment group, treatment day, and study day by treatment interaction, with baseline measured at each study day as a covariate; Mean Difference (Final Values) = 25.02, 95% CI 2-sided [16.10 to 33.94], Standard Error of Mean 4.52

2. Secondary Outcome: Baseline Adjusted Peak Expiratory Flow (PEF) Area Under The Concentration Time Curve Up From Time Zero up to 6 Hours (AUC0-6) Over 3 Weeks
Description: Serial PEF measurements were obtained via spirometry. PEF measures for purpose of serial PEF assessment (pre and postdose) were collected from the spirometer assessed PEF, utilizing the values from the efforts selected based on the highest of 3 acceptable FEV1 maneuvers.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters/min*hour
Arm/Group | Placebo MDPI QID | Albuterol MDPI 180 mcg QID
Number analyzed (Participants) | 92 | 92
Liters/min*hour | 71.52 (10.201) | 147.85 (10.245)
Statistical Analysis 1: Comparison: Placebo MDPI QID vs Albuterol MDPI 180 mcg QID; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 76.33, 95% CI 2-sided [47.76 to 104.91], Standard Error of Mean 14.47

3. Secondary Outcome: Summary of Participants With Adverse Events
Description: Adverse events (AEs) summarized in this table are those that began or worsened after treatment with study drug (treatment-emergent AEs). An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator as mild (no limitation of usual activities), moderate, or severe (inability to carry out usual activities).
  Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: 6 Months
Population: Safety Analysis set includes all participants who receive at least 1 dose of study drug. In this population, treatment is assigned based upon the treatment participants actually receive, regardless of the treatment to which they were randomized.
Measure: Number; unit: participants
Arm/Group | Placebo MDPI QID | Albuterol MDPI 180 mcg QID
Number analyzed (Participants) | 92 | 93
participants
  Any adverse event | 21 | 21
  Severe adverse event | 0 | 0
  Treatment-related adverse event | 0 | 0
  Deaths | 0 | 0
  Other serious AE | 0 | 0
  Withdrawn from study due to AE | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 22
Arm/Group | Placebo MDPI QID | Albuterol MDPI 180 mcg QID
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/93
Other Adverse Events (participants affected / at risk) | 19/92 | 9/93
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo MDPI QID (N=92) | Albuterol MDPI 180 mcg QID (N=93)
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3
Pyrexia (General disorders) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 0
Headache (Nervous system disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.